Evaluation of Delefilcon A and Senofilcon A Daily Disposable Toric Soft Contact Lenses Over Two Weeks of Wear

Protocol CR-6553

Version: 3.0

Date: 27 November 2023

Investigational Products: The Test product will be rotationally stabilized, astigmatic, soft contact lenses in senofilcon A with a chromophore to filter High-Energy Visible Light (HEVL). The Control product will be Alcon DAILIES TOTAL1® for Astigmatism Daily Contact Lenses (DT1fA).

Keywords: Astigmatism, toric contact lenses, senofilcon A, RTY-1 chromophore, High-Energy Visible Light, Alcon DAILIES TOTAL1® for Astigmatism, delefilcon A, daily wear, daily disposable, dispensing, Single use Eye-Cept® Rewetting Drops, LacriPure Saline Solution, ScleralFil Preservative Free Saline Solution, CLUE comfort, CLUE vision, CLUE handling, logMAR visual acuity, rotational performance.

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This clinical trial will be conducted in compliance with ISO 14155:2020 Clinical investigation of medical devices for human subjects – Good clinical practice<sup>1</sup> and the Declaration of Helsinki.<sup>2</sup>

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

#### TABLE OF CONTENTS

| PF | ROT | OCOL TITLE, NUMBER, VERSION AND DATE | 6 |
|----|------|-------------------------------------------------------------|----|
| | | SOR NAME AND ADDRESS | |
| M | EDI | CAL MONITOR | 6 |
| ΑÌ | UTH | ORIZED SIGNATURES | 7 |
| CI | HAN | IGE HISTORY | 8 |
| S | γNΟ | PSIS | 9 |
| C | OMN | MONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS | 14 |
| 1. | | NTRODUCTION AND BACKGROUND | |
| | 1.1. | Name and Descriptions of Investigational Products | 15 |
| | 1.2. | Intended Use of Investigational Products | 15 |
| | 1.3. | | |
| | 1.4. | Summary of Known Risks and Benefits to Human Subjects | 15 |
| | 1.5. | | |
| 2. | 5 | STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 16 |
| | 2.1. | | |
| | 2.2. | Endpoints | 16 |
| | 2.3. | Hypotheses | 17 |
| 3. | - | FARGETED STUDY POPULATION | 17 |
| | 3.1. | General Characteristics | 17 |
| | 3.2. | Inclusion Criteria | 17 |
| | 3.3. | Exclusion Criteria | 18 |
| | 3.4. | Enrollment Strategy | 18 |
| 4. | 5 | STUDY DESIGN AND RATIONALE | 18 |
| | 4.1. | Description of Study Design | 18 |
| | 4.2. | Study Design Rationale | 19 |
| | 4.3. | Enrollment Target and Study Duration | 19 |
| 5. | - | FEST ARTICLE ALLOCATION AND MASKING | 19 |
| | 5.1. | Test Article Allocation | 19 |
| | 5.2. | Masking | 20 |
| | 5.3. | Procedures for Maintaining and Breaking the Masking | 20 |
| 6. | 5 | STUDY INTERVENTION | 20 |
| | 6.1. | Identity of Test Articles | 20 |
| | 6.2. | Ancillary Supplies/Products | 21 |
| | 6.3. | Administration of Test Articles | 22 |
| | 6.4. | Packaging and Labeling | 22 |
| | 6.5. | Storage Conditions | 22 |
| | 6.6. | Collection and Storage of Samples | 22 |

| ( | 5.7. | Accountability of Test Articles | 22 |
|---|---|---|---|
| 7. | STU | JDY EVALUATIONS | 23 |
| , | 7.1. | Time and Event Schedule | 23 |
| , | 7.2. | Detailed Study Procedures | 25 |
| | VIS | SIT 1 | 25 |
| | VIS | SIT 2 | 31 |
| | VIS | NT 3 | 33 |
| | VIS | SIT 4 | 35 |
| | VIS | SIT 5 | 35 |
| | VIS | SIT 6 | 35 |
| | FIN | AL EVALUATION | 37 |
| , | 7.3. | Unscheduled Visits | 37 |
| , | 7.4. | Laboratory Procedures | 38 |
| 8. | SU | BJECTS COMPLETION/WITHDRAWAL | 39 |
| 8 | 8.1. | Completion Criteria | 39 |
| 8 | 8.2. | Withdrawal/Discontinuation from the Study | 39 |
| 9. | PRI | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 39 |
| ( | 9.1. | Systemic Medications | 39 |
| 10. | DE | VIATIONS FROM THE PROTOCOL | 40 |
| 11. | STU | JDY TERMINATION | 41 |
| 12. | PRO | OCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 42 |
| 13. | AD | VERSE EVENTS | 43 |
| | 13.1. | Definitions and Classifications | 43 |
| | 13.2. | Assessing Adverse Events | 44 |
| | 13.2 | 2.1. Causality Assessment | 45 |
| | 13.2 | 2.2. Severity Assessment | 45 |
| | 13.3. | Documentation and Follow-Up of Adverse Events | 45 |
| | 13.4. | Reporting Adverse Events | |
| | 13.4 | 4.1. Reporting Adverse Events to Sponsor | 46 |
| | 13.4 | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities | 47 |
| | 13.5. | Event of Special Interest | |
| | 13.6. | Reporting of Pregnancy | 47 |
| 14. | STA | ATISTICAL METHODS | 48 |
| | 14.1. | General Considerations | 48 |
| | 14.2. | Sample Size Justification | |
| | 14.3. | Analysis Populations | |
| | 14.4. | Level of Statistical Significance. | |
| | 14.5. | Primary Analysis | 49 |

| 14.6. | Secondary Analysis | 49 |
|---|---|---|
| 14.7. | Exploratory Analyses | 49 |
| 14.8. | Interim Analysis | 50 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 50 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 50 |
| 15. DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 50 |
| 15.1. | Electronic Case Report Form/Data Collection | 50 |
| 15.2. | Subject Record | 51 |
| 15.3. | Trial Registration on ClinicalTrials.gov | 51 |
| 16. DA | TA MANAGEMENT | 51 |
| 16.1. | Access to Source Data/Document | 51 |
| 16.2. | Confidentiality of Information | 51 |
| 16.3. | Data Quality Assurance | 51 |
| 16.4. | Data Monitoring Committee (DMC) | 52 |
| 17. CL | INICAL MONITORING | 52 |
| 18. ET | HICAL AND REGULATORY ASPECTS | 52 |
| 18.1. | Study-Specific Design Considerations | 52 |
| 18.2. | Investigator Responsibility | 52 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 53 |
| 18.4. | Informed Consent | 53 |
| 18.5. | Privacy of Personal Data | 54 |
| 19. ST | UDY RECORD RETENTION | 55 |
| 20. FIN | NANCIAL CONSIDERATIONS | 55 |
| 21. PU | BLICATION | 55 |
| 22. RE | FERENCES | 55 |
| APPEND | OIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 57 |
| APPEND | OIX B: PATIENT INSTRUCTION GUIDE | 79 |
| APPEND | DIX C: PACKAGE INSERT (APPROVED PRODUCT) | 80 |
| APPEND | <u></u> | |
| | LENS FITTING CHARACTERISTICS | |
| | SUBJECT REPORTED OCULAR SYMPTOMS | 90 |
| | DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS | 92 |
| | BIOMICROSCOPY SCALE | 98 |
| | DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION | 104 |
| | TORIC FIT EVALUATION | |
| | DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE | |
| | PATIENT REPORTED OUTCOMES | |
| | LENS INSERTION AND REMOVAL | |

| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING | 123 |
|---|---|
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 132 |
| LIST OF TABLES | |
| Table 1: Test Articles | 21 |
| Table 2: Ancillary Supplies | 21 |
| Table 3: Time and Events | 23 |
| Table 4: Disallowed systemic medications. | 40 |
| Table 5: Disallowed systemic antihistamines | 40 |
| Table 6: Examples of major and minor protocol deviations | 41 |
| Table 7: Half-Width of the 95% Confidence Intervals for Proportion of Eyes with Grade 3+ SLFs | 48 |
| LIST OF FIGURES | |
| Figure 1: Study Flowchart | 13 |

#### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Evaluation of Delefilcon A and Senofilcon A Daily Disposable Toric Soft Contact Lenses Over Two Weeks

of Wear

Protocol Number: CR-6553

Version: 3.0

Date: 27 November 2023

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, <sup>3</sup> ISO 14155:2020, <sup>1</sup> and the Declaration of Helsinki. <sup>2</sup>

| Author & Study | Con Floritonia Simulatura Portuga | |
|-----------------------|-----------------------------------|------|
| Responsible Clinician | See Electronic Signature Report | DATE |
| Medical Monitor | See Electronic Signature Report | |
| | | DATE |
| Clinical Operations | | |
| Manager | See Electronic Signature Report | |
| | | DATE |
| Biostatistician | See Electronic Signature Report | |
| | | DATE |
| Data Management | See Electronic Signature Report | |
| | | DATE |
| Medical Safety | | |
| Officer | See Electronic Signature Report | - |
| | | DATE |
| Approver | See Electronic Signature Report | 15 |
| | | DATE |

### CHANGE HISTORY

| Version | Originator | Description of Change(s) and<br>Section Number(s) Affected | Justification for Change | Date | |
|---|---|---|---|---|---|
| 1.0 | | Original Protocol | N/A | 10<br>2023 | OCT |
| 2.0 | | Minor corrections to wording for PRO items in PRO spec (Appendix A) | Minor errors in PRO item wording | 09<br>2023 | NOV |
| 3.0 | | The following changes were made in Section 7.2 – Detailed Study Procedures: 1. Corrected sentences describing the order of PRO questionnaires for baseline and follow-up visits (study procedure steps 1.8, 2.4, 3.5, 6.5). 2. Removed incorrect sentence under Visit 5 of detailed study procedures that instructed subjects to bring habitual spectacles or contact lenses to this visit. 3. Updated lens dispensing instructions (steps 1.29, 2.13) to clarify that the return window requirement holds regardless of whether the dispensing and/or follow-up visit days are counted toward the minimum wear requirement. | questionnaires was incorrectly described for the baseline and follow-up visits. 2. Unnecessary to bring habitual correction to visit 5 as study lens wear will continue following this visit. 3. Lens dispensing instructions updated for clarity. | 27 2023 | NOV |

#### **SYNOPSIS**

| Evaluation of Delefilcon A and Senofilcon A Daily Disposable Torio |
|---|
| Contact Lenses Over Two Weeks of Wear |
| JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 Clinical Trial Phase: Confirmatory |
| Design control phase: Confirmatory phase, phase 3 |
| This study will be registered on ClinicalTrials.gov by the Sponsor. Investigational Product (Test lens): The test product will be rotationally |
| stabilized astigmatic soft contact lenses in senofilcon A with a chromophor to filter High-Energy Visible Light (HEVL). Approved Product (Control lens): The control product will be DAILIE TOTAL1® for Astigmatism Contact Lenses (DT1fA). |
| Wear Schedule: Daily wear |
| Replacement Schedule: Daily disposable |
| Primary Objective: The primary objective of this study is to estimate the incidence rate (percentage) of eyes with clinically significant slit-lamp findings (Grade 3 or 4) related to each study lens (Test lens and Control lens) after approximately 2-weeks of lens wear. |
| Exploratory Objectives: The exploratory objectives of this study include the estimation of the mean difference between study lenses (Test lens and Control lens) with respect to distance monocular high luminance, high contrast (HLHC), logMAR visual acuity (at the 1-week follow-up visit), and CLUE comfort, vision, and handling scores (at the fitting, 1- and 2-week follow-up visits). Additional exploratory objectives of the study are to estimate the mean and standard deviation of the mean settled toric orientation of each study lens (Test lens and Control lens) following lens settling and after 1- and 2-weeks of lens wear, and to assess the toric lens orientation of each study lens, 1- and 3-minutes after lens insertion. Adverse events will also be monitored and collected. |
| <ul> <li>Primary endpoint: <ul> <li>Indicidence (percentage) of eyes with Grade 3 or 4 slit lamp findings related to the study lenses (Test lens and Control lens) after 2-week of lens wear.</li> </ul> </li> <li>Exploratory endpoints: <ul> <li>Distance Monocular HLHC logMAR at 4m at the 1-week follow-up visit</li> <li>Contact Lens User Experience (CLUE) comfort scores at the fitting, 1-, and 2-week follow-up visits</li> <li>CLUE vision scores at the fitting, 1-, and 2-week follow-up visits</li> <li>CLUE handling scores at the fitting, 1-, and 2-week follow-up visits</li> </ul> </li> <li>Lens orientation at 1 minute and 3 minutes following insertion at fitting</li> <li>Mean Settled Lens Orientation at the fitting, 1-, and 2-week follow-up visits</li> </ul> |

| Study Design | This will be a multi-site, bilateral, dispensing, randomized, controlled, double-masked, 2×2 crossover study. Eligible subjects will be randomly assigned to one of two lens wear sequences (Test/Control or Control/Test). Each lens will be worn for a period of 14(±4) days. There will be a 7(±2) days washout period between study lenses. There will be a total of 6 visits: Visit 1: Screening, baseline evaluation and lens fit #1 Visit 2: Follow-up evaluation #1 (for first lens dispensed) Visit 3: Follow-up evaluation #2 (for first lens dispensed) Visit 4: Continuance, lens fit #2 Visit 5: Follow-up evaluation #3 (for second lens dispensed) Visit 6: Follow-up evaluation #4 (for second lens dispensed) See the flow chart at the end of the synopsis table for a schematic of the |
|---|---|
| Sample Size | study visits and procedures (Figure 1). This study will have an enrollment target of approximately 66 subjects, with |
| Sample Size | a target of at least 60 to complete (assuming a dropout rate of 10%). |
| Study Duration | Total study duration including the enrollment period is anticipated to be approximately 10 weeks. |
| Anticipated Study Population | Subjects will be habitual soft contact lens wearers with bilateral astigmatism who are between 18 and 39 years of age (inclusive). |
| Eligibility Criteria - Inclusion | Potential subjects must satisfy of all the following criteria to be enrolled in |
| | Inclusion Criteria following Screening The subject must: 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form. 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol. 3. Be between 18 and 39 (inclusive) years of age at the time of screening. 4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past four weeks. 5. Possess a wearable pair of spectacles that provide correction for distance vision. Inclusion Criteria at Baseline Evaluation The subject must: 6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study: a. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps b. Cylinder powers (DC) -0.75 and -1.25 c. Axes (°) 170, 180, 10, 80, 90, 100 7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye. |

| Eligibility Criteria – Exclusion | Potential subjects who meet any of the following criteria will be excluded from participating in the study: |
|---|---|
| | Exclusion Criteria following Screening The subject must not: |
| | 1. Be currently pregnant or lactating. |
| | <ul><li>2. Be diabetic.</li><li>3. Be currently using any ocular medications or have any ocular infection</li></ul> |
| | of any type. |
| | <ol> <li>By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.</li> <li>Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.</li> <li>Be currently wearing monovision or multifocal contact lenses.</li> <li>Be currently wearing lenses in an extended wear modality.</li> <li>Have a history of strabismus or amblyopia.</li> <li>Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.</li> <li>Have participated in a contact lens or lens care product clinical trial</li> </ol> |
| | within 7 days prior to study enrollment. |
| | Exclusion Criteria at Baseline Evaluation |
| | The subject must not: |
| | 11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). |
| | 12. Have fluctuations in vision due to clinically significant dry eye or other |
| | ocular conditions. |
| | 13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.). |
| Disallowed | Subjects will not be eligible to enroll if they are taking any ocular |
| Medications/Interventions | medications, or any systemic medications that would normally contraindicate contact lens wear or may otherwise compromise study endpoints. See section 9.1 for details regarding disallowed systemic medications. |

| Measurements and Procedures | The key procedures associated with the endpoints for this study will be: |
|---|---|
| 110000010110110001100000000000000000000 | - Examination of the anterior segment using a slit lamp biomicroscope and grading findings using the FDA grading scale |
| | - Measurement of HLHC VA using ETDRS charts |
| | - Measurement of toric lens orientation and rotational stability using a slit |
| | lamp biomicroscope |
| | - Overseeing completion of the CLUE questionnaires |
| Microbiology or Other | Not applicable for this study. |
| Laboratory Testing | |
| Study Termination | The occurrence of an Unanticipated Adverse Device Effect (UADE) or |
| | Serious Adverse Event (SAE) for which a causal relationship to a test article |
| | cannot be ruled out, will result in stopping further dispensing investigational |
| | product. In the event of a UADE or SAE, the Sponsor Medical Monitor may |
| | unmask the treatment regimen of subject(s) and may discuss this with the |
| | Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- Lens cases, fluorescein strips and preservative-free rewetting dr | |
| Specific Materials | artificial tears will be supplied for use as needed. |
| Principal Investigator(s) and A full list of Principal Investigators, clinical sites, and institutions | |
| Study Institution(s)/Site(s) separately from the Study Protocol and is included in the study | |
| | File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADE Adverse Device Effect

ADHD Attention Deficit Hyperactivity Disorder
AE Adverse Event/Adverse Experience
BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience
COM Clinical Operations Manager
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

D Diopter

DMC Data Monitoring Committee
eCRF Electronic Case Report Form
EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration GCP Good Clinical Practice HEVL High Energy Visible Light

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure

ICH The International Council for Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LASIK Laser-Assisted in Situ Keratomileusis

LogMAR Logarithm of Minimal Angle of Resolution

OD Right Eye
OS Left Eye
OU Both Eyes

PIG Patient Instruction Guide
PQC Product Quality Complaint
PRK Photorefractive Keratectomy
PRO Patient Reported Outcome

QA Quality Assurance

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan
SAS Statistical Analysis System
SD Standard Deviation
SLF Slit Lamp Finding

UADE Unanticipated Adverse Device Effect
USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

DAILIES TOTAL1® for Astigmatism Contact Lenses (DT1fA) are single-use, daily disposable lenses indicated for the correction of astigmatism and associated ametropia in persons with non-diseased eyes. The purpose of this study is to evaluate the ocular physiological response following wear of a daily disposable, toric lens design in senofilcon A incorporating a HEVL-filtering chromophore (RTY-1) relative to DT1fA as Control.

#### 1.1. Name and Descriptions of Investigational Products

The Test lens in this study will be a toric contact lens design in senofilcon A containing a HEVL-filtering chromophore (RTY-1).

The Control lens in this study will be DT1fA. DT1fA contact lenses are made from a lens material that is 33% water and 67% (delefilcon A) polymer, a silicone containing hydrogel with added phosphatidylcholine. DT1fA lenses also contain a handling tint (color additive copper phthalocyanine).

Further details about the Test and Control articles are found in section 6.1 of this protocol, the Investigator's Brochure<sup>4</sup> and in the DT1fA package insert (Appendix C).

#### 1.2. Intended Use of Investigational Products

The intended use of the investigational products is the correction of astigmatism and associated myopic refractive error. Study lenses will be worn bilaterally in a daily wear, daily disposable modality for at least 8 hours per day. Each wear period will be 14±4 (i.e., 10 to 18) days in duration, and subjects will be instructed to wear lenses for at least 5 days per week during each wear period. Two wear periods will be completed, with a washout period of 7±2 days between the wear periods.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings for the test lens were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding the test design refer to the Investigator's Brochure.<sup>4</sup>

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The anticipated clinical benefit of the investigational lenses will be the correction of refractive error. No adverse device effects are anticipated. The risks associated with use of the investigational lenses are considered to be the same as those for other marketed soft contact lens worn in the same modality (i.e., daily disposable wear). No additional risks associated with participation in this investigation are anticipated.

Comprehensive risk and benefit information regarding the investigational (test lens) design and the DT1fA control lens are included in the Investigator's Brochure<sup>4</sup> and the DT1fA package insert (Appendix C), respectively.

#### 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Prototype toric lens designs featuring the RTY-1 chromophore have previously been evaluated in several JJVC-sponsored clinical trials. Safety data from these trials suggest the investigational lenses have a safety profile equivalent to currently marketed soft contact lens products; a review of literature references and prior clinical data related to the test designs is given in the Investigator's Brochure.<sup>4</sup>

DT1fA contact lenses are approved in the US for the correction of astigmatism and associated ametropia in persons with non-diseased eyes. For further details regarding the DT1fA control lens, refer to the DT1fA package insert (Appendix C).


#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

#### Primary Objective:

The primary objective of this study is to estimate the incidence rate (percentage) of eyes with clinically significant slit-lamp findings (Grade 3 or 4) related to each study lens (Test lens and Control lens) after approximately 2-weeks of lens wear.

#### **Exploratory Objectives:**

The exploratory objectives of this study include the estimation of the mean difference between study lenses (Test lens and Control lens) with respect to distance monocular high luminance, high contrast (HLHC), logMAR visual acuity (at the 1-week follow-up visit), and CLUE comfort, vision, and handling scores (at the fitting, 1- and 2-week follow-up visits). Additional exploratory objectives of the study are to estimate the mean and standard deviation of the settled toric roation of each study lens (Test lens and Control lens) following lens settling and after 1- and 2-weeks of lens wear, and to assess the toric lens orientation of each study lens, 1- and 3-minutes after lens insertion. Adverse events will also be monitored and collected.

#### 2.2. Endpoints

#### Primary endpoint:

#### 1. Percentage of Eyes with slit-lamp findings (Grade 3 or 4) related to study lens wear

Slit Lamp Findings (Grade 3 or higher) will be assessed for each subject eye at all study visits (scheduled and unscheduled). However, the primary endpoint will be the percentage of eyes with Grade 3 or higher SLFs related to study lens wear, after approximately 2 weeks of lens wear.

SLFs will be evaluated and classified using the FDA Grading scale rating from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e., Grade 1=trace, Grade 2= mild, Grade 3=moderate and Grade 4= severe).

#### **Exploratory Endpoints:**

#### 1. Distance Monocular HLHC logMAR Visual Acuity

Visual acuity (VA) will be assessed monocularly at the 1-week follow-up visits under high-luminance high contrast (HLHC) conditions at a test distance of 4 meters using ETDRS Charts. The logMAR VA score is a continuous endpoint.

#### 2. CLUE Comfort Scores

Subjective comfort will be assessed using the Contact Lens User Experience (CLUE) questionnaire. CLUE will be assessed at the fitting, 1- and 2-week follow-up visits. The CLUE comfort score is a conintuous endpoint.

CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>TM</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>TM</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>5</sup>

- 3. <u>CLUE Vision Scores</u> at the fitting, 1-, and 2-week follow-up visits. The CLUE vision score is a conintuous endpoint.
- 4. <u>CLUE Handling Scores</u> at the fitting, 1-, and 2-week follow-up visits. The CLUE handling score is a conintuous endpoint.


#### 5. Toric Lens Orientation

Toric lens orientation (scribe mark position relative to 6 o'clock) will be assessed for each eye at 1, 3 and at least 15 minutes after lens insertion at the fitting visit, and at the 1- and 2-week follow-up visits. However, toric lens orientation at 1- and 3-minutes after lens insertion at the fitting visit is the exploratory endpoint. The endpoint is the distribution (counts, percentages) of eyes for the toric Orientation (in degrees).

#### 6. Mean Settled Lens Orientation

Lens orientation (scribe mark position relative to 6 o'clock) will be assessed for each eye at 1 minute, 3 minutes, at least 15 minutes after lens insertion; 2 additional measurements per eye following settling will also be collected. The exploratory endpoint is the lens orientation assessed at the fitting, 1-, and 2-week follow-up visits. Mean settled lens orientation is a continuous response where the mean is calculated by eye by averaging across all lens orientation measurements collected at least 15-minutes after lens insertion. The standard deviation of average settled lens orientation will also be calculated. See in Appendix D for details regarding the collection of lens orientation.

7. Adverse events (AEs) - including ocular and non-ocular. Details for AEs will be provided through listings.

#### 2.3. Hypotheses

Not applicable, there is no planned hypothesis testing for any endpoints in this study.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

The target population for this study will be healthy adult soft contact lens wearers between 18 and 39 years of age with binocular myopic astigmatism.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

Inclusion Criteria following Screening

The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be between 18 and 39 (inclusive) years of age at the time of screening.
- 4. By self-report, habitually wear soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e., not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 2 days per week during the past four weeks.
- 5. Possess a wearable pair of spectacles that provide correction for distance vision.

Inclusion Criteria at Baseline Evaluation

The subject must:

- 6. In both eyes, have refractive error suitable for correction with the toric contact lens powers available in this study:
  - a. Sphere powers (DS) -1.50 through -4.00 in 0.25 steps
  - b. Cylinder powers (DC) -0.75 and -1.25
  - c. Axes (°) 170, 180, 10, 80, 90, 100

7. Have best corrected monocular distance visual acuity of 20/30 or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria following Screening

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Be diabetic.
- 3. Be currently using any ocular medications or have any ocular infection of any type.
- 4. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g., rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
- 5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
- 6. Be currently wearing monovision or multifocal contact lenses.
- 7. Be currently wearing lenses in an extended wear modality.
- 8. Have a history of strabismus or amblyopia.
- 9. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
- 10. Have participated in a contact lens or lens care product clinical trial within 7 days prior to study enrollment.

Exclusion Criteria at Baseline Evaluation

The subject must not:

- 11. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
- 12. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
- 13. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This will be a mulit-site, 6-visit, randomized, controlled, double-masked, bilateral wear, dispensing 2×2 crossover study.

At the initial visit (Visit 1), if a subject is deemed eligible, the subject will be randomized into one of two unique sequences of lens wear (Test/Control or Control/Test), otherwise, the subject will be deemed ineligible and exited from the study.


Subjects will wear each study lens (Test lens and Control lens) in a daily wear, daily disposable modality for approximately 2 weeks. There will be a washout period of 7±2 days between wear periods. Subjects will not have access to the study lenses following completion of the protocol.

Subjects will be advised to wear the study lenses for a minimum of 8 hours per day for at least 5 days during each wear period. Unscheduled visits may be conducted, if appropriate, and lost or damaged lenses may be replaced when necessary.

#### 4.2. Study Design Rationale

A 6-visit, double-masked,  $2\times2$  crossover study design was chosen to demonstrate the study objectives. In this design, each subject will act as their own control to reduce the influence of potential confounding factors such as age, gender, race, and vision correction. To help further reduce the potential for carryover effects, a washout period of approximately 1-week ( $7\pm2$  days) between study will be used.

#### 4.3. Enrollment Target and Study Duration

This study will have an enrollment target of approximately 66 subjects, with a target of at least 60 to complete. The study will be conducted at up to 6 clinical sites, where the enrollment target for each site will be approximately 11 subjects. A subject will be considered enrolled upon signing of the informed consent form.

There will be 6 visits in total per subject. The total study duration including the enrollment period is expected to be approximately 10 weeks. Subjects who are discontinued prior to the final evaluation may be replaced at the discretion of the study sponsor. The investigation will end at the time that the study data is hard locked.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn bilaterally in a randomized fashion using a 2×2 crossover design with 2 lens types and 2 periods.

A computer-generated randomization scheme will be used to randomly assign subjects to one of two unique sequences of lens wear. The randomization scheme will be provided by an internal independent unmasked Biostatistician who is independent of the study team and not involved in the study conduct or analyses, beyond the randomization codes and schedule generation. The randomization scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).

The assignment of subjects will be performed at the first visit prior to the first fitting. Clinical sites must follow the randomization scheme provided. The following must have occurred prior to randomization:

- Informed consent must have been obtained
- The subject must have met all inclusion and exclusion criteria
- The subject history and baseline information must have been collected

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the randomization scheme (lens fitting schedule) to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme (lens fitting schedule).
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.


#### 5.2. Masking

To reduce the possibility of bias, this will be a double-masked trial. Subjects and investigators and clinical site personel will not be aware of the identity of the assigned lenses. While every effort will be made to maintain masking of study investigators, due to differences in the lens designs, it is possible that investigators may determine the identity of the designs during study procedures.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Every attempt will be made to keep the clinical trial personnel involved in the study (e.g., data management, project biostatistician, and clinical operations) unaware of the identity of the assigned study lenses. The identity of the study lenses will be masked by having the blister packs labeled with the study number, lot number, sphere power, cylinder power, axis, expiration date, and randomization code. During study execution, only the independent unmasked biostatistician generating the lens fitting schedule will have access to the decode information that allows matching of the randomization codes to the test articles. The medical monitor will also have access to the decode information in case breaking the mask is necessary for the urgent medical treatment of a subject. All personnel involved in the study will be unmasked once the study database is locked.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced at the discretion of the study sponsor.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test | Control |
|---|---|---|
| Test Article Form | Soft con | tact lens |
| Brand and Product Name | TRA1xx and TRA2xx series toric<br>contact lens with HEVL-filtering<br>chromophore | DAILIES TOTAL1® for<br>Astigmatism |
| Manufacturer | Johnson & Johnson Vision Care,<br>Inc. | Alcon Laboratories, Inc. |
| Packaging Form | Blister packaging in s | terile packing solution |
| Packaging Solution | Optimized Borate Buffer (OBB) solution | Phosphate buffered saline solution with wetting agents |
| Lens Material | senofilcon A (C3) with RTY-1<br>chromophore | delefilcon A |
| Sphere Powers (DS) | -1.50 to -4.00 in 0.25 steps | |
| Cylinder Powers (DC) | -0.75, -1.25 | |
| Cylinder Axes (°) | 10, 80, 90, 100, 170, 180 | |
| Nominal Water Content (%) | 38% | 33% |
| Nominal Base Curve (mm) | 8.5 | 8.6 |
| Lens Diameter (mm) | 14.3 | 14.5 |
| Fiducial marks | 6 and 12 o'clock fiducial lines | 6 o'clock scribe mark |
| Dk (intrinsic Dk-Coulometric method, ×10-11 [cm2 /sec] [ml O2/ml × mm Hg] at 35°C) | 103 | 140 |
| Modality in Current Study | Daily wear | |
| Replacement Frequency in<br>Current Study | Daily di | sposable |

In total, both Test and Control lenses will be available in 132 unique lens powers (11 sphere powers  $\times$  2 cylinder powers  $\times$  6 axes).

The total number of test lenses to be used in this study (not including lenses that are replaced due to droppage, loss or damage) is expected to be approximately 1848 lenses (target enrollment of 66 subjects  $\times$  2 eyes per subject  $\times$  14 day wear period). Test and Control lenses will be worn in a 1:1 ratio, thus the number of control lenses to be used is expected to be approximately the same (1848 lenses).

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Non-Preserved Rewetting Drops | | |
|---|---|---|---|
| Solution Name/Description | Single use Eye-Cept® | LacriPure Saline | ScleralFil Preservative |
| Solution Name/Description | Rewetting Drops | Solution | Free Saline Solution |
| Manufacturer | Optics Laboratory | Menicon | Bausch & Lomb |
| Preservative | None | None | None |

Lens cases and fluorescein strips (either 0.6 mg or 1.0 mg) will be supplied for use as needed.

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the investigator and/or the sponsor.

#### 6.4. Packaging and Labeling

The test articles will be supplied in blister packages as the primary packaging and placed into plastic bags as secondary packaging. Test and Control blister packages will be physically over-labeled with permanent labels. Representative sample labels for the primary and secondary packaging are shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

No samples will be collected as part of the study procedures. When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted for. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject-returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Lens Fitting<br>#1 | Visit 2<br>Follow-up<br>#1 | Visit 3<br>Follow-up<br>#2 | Visit 4<br>Continuanc<br>e, Lens<br>Fitting #2 | Visit 5<br>Follow-up<br>#3 | Visit 6<br>Follow-up<br>#4, Final<br>Evaluation |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | 7 ± 2 days<br>following<br>Visit 1 | 7 ± 2 days<br>following<br>Visit 2 | 7 ± 2 days<br>following<br>Visit 3 | 7 ± 2 days<br>following<br>Visit 4 | 7 ± 2 days<br>following<br>Visit 5 |
| Minimum lens<br>wear time<br>immediately prior<br>to visit | Must wear<br>habitual<br>lenses | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) | No<br>requirement<br>for this visit | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) |
| Estimated Visit<br>Duration | 2.5 hours | 1.5 hours | 1 hour | 1.5 hours | 1.5 hours | 1 hour |
| Statement of informed consent | x | | | | | |
| Demographics | X | 54 | | | | |
| Medical history<br>and concomitant<br>medications | x | х | х | x | х | x |
| Habitual contact<br>lens information | x | | | | | |
| Habitual lens wear time | x | | | | | |
| Eligibility at<br>Screening | x | | | | | |
| Subject reported ocular symptoms | x | x | x | x | x | x |
| Baseline PRO<br>questionnaire | x | | | | | 5 |
| Entrance visual acuity | x | х | x | x | x | х |
| Remove habitual lenses | x | | | x | | |

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Lens Fitting<br>#1 | Visit 2<br>Follow-up<br>#1 | Visit 3<br>Follow-up<br>#2 | Visit 4<br>Continuanc<br>e, Lens<br>Fitting #2 | Visit 5<br>Follow-up<br>#3 | Visit 6<br>Follow-up<br>#4, Final<br>Evaluation |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | 7 ± 2 days<br>following<br>Visit 1 | 7 ± 2 days<br>following<br>Visit 2 | 7 ± 2 days<br>following<br>Visit 3 | 7 ± 2 days<br>following<br>Visit 4 | 7 ± 2 days<br>following<br>Visit 5 |
| Minimum lens<br>wear time<br>immediately prior<br>to visit | Must wear<br>habitual<br>lenses | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) | No<br>requirement<br>for this visit | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) |
| Estimated Visit<br>Duration | 2.5 hours | 1.5 hours | 1 hour | 1.5 hours | 1.5 hours | 1 hour |
| Subjective Sphero-<br>Cylindrical<br>Refraction | x | | | | | x |
| Slit Lamp<br>Biomicroscopy | x | X | x | x | x | X |
| Eligibility at<br>Baseline | x | | | | | |
| Lens Selection | X | | | X | | |
| Lens insertion and<br>timed rotation<br>assessments | x | | | x | | |
| Lens settling | x | | | x | | |
| Toric fit assessment | x | | 3 | x | | |
| General fit<br>assessment | x | | | x | | |
| Spherical over-<br>refraction | x | A. | | x | | |
| Lens modification<br>(if necessary) | x | | | x | | |
| Post-fit PRO<br>questionnaire | x | | | x | | |
| Additional samples<br>of toric lens<br>orientation<br>(performed twice) | х | | x | x | | х |
| Exit visual acuity | X | X | X | X | X | |
| Dispensing criteria | x | 9 | * | X | V V | 9 |
| Dispensing instructions | x | x | | x | x | |
| Schedule next visit | X | X | X | X | Х | |
| Wear time and compliance | | х | x | | x | x |
| Collect unworn<br>lenses | | 0.00 | x | | | x |
| Follow-up PRO questionnaire | | x | x | | x | x |
| Distance HLHC<br>visual acuity using<br>ETDRS charts | | х | | | Х | |

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Lens Fitting<br>#1 | Visit 2<br>Follow-up<br>#1 | Visit 3<br>Follow-up<br>#2 | Visit 4<br>Continuanc<br>e, Lens<br>Fitting #2 | Visit 5<br>Follow-up<br>#3 | Visit 6<br>Follow-up<br>#4, Final<br>Evaluation |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | 7 ± 2 days<br>following<br>Visit 1 | 7 ± 2 days<br>following<br>Visit 2 | 7 ± 2 days<br>following<br>Visit 3 | 7 ± 2 days<br>following<br>Visit 4 | 7 ± 2 days<br>following<br>Visit 5 |
| Minimum lens<br>wear time<br>immediately prior<br>to visit | Must wear<br>habitual<br>lenses | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) | No<br>requirement<br>for this visit | 1 hour<br>(study<br>lenses) | 1 hour<br>(study<br>lenses) |
| Estimated Visit<br>Duration | 2.5 hours | 1.5 hours | 1 hour | 1.5 hours | 1.5 hours | 1 hour |
| Toric lens<br>orientation | | x | x | | x | x |
| Lens removal | | X | X | | X | X |
| Lens reinsertion and settling | | x | | | x | |
| Continuance | | | | х | | |
| Subject completion status | | | | | | X |

#### 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must wear their habitual contact lenses to this visit.

| | | Visit 1: Screening |
|---|---|---|
| Step | Procedure | Details |
| 1.1. | Statement of Informed<br>Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2. | Demographics | Record the subject's year of birth, age, gender, race and ethnicity. |
| 1.3. | Medical History and<br>Concomitant<br>Medications | Record the subject's medical history and concomitant medications. |
| 1.4. | Habitual Lenses | Record the subject's habitual lens type, parameters, lens care solution, wear modality, and approximate prescription date. |
| 1.5. | Habitual lens wear time. | Record the average and comfortable wear time for the subject's habitual contact lenses. |

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.6. | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |
| | | If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms do not need to be completed as part of Final Evaluation. |

| | | Visit 1: Baseline | <u> </u> |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.7. | Subject reported ocular symptoms | Record any subject reported ocular symptoms reported with regard to their habitual contact lenses. | 552 |
| 1.8. | Baseline PRO questionnaire | Ask the subject to fill out the baseline questionnaire regarding their experience with their habitual contact lenses. The glare PRO questionnaire will be completed first, | |
| 1.9. | Entrance visual acuity | followed by the CLUE questionnaire, followed by the other PRO items. Record the monocular distance Snellen visual acuity for each eye (OD, OS) to the nearest letter with the subject's habitual contact lens correction. Subjects must continue until at least 50% of the letters on a line | |
| 1.10. | Remove habitual lenses | are read incorrectly. The subject's habitual contact lenses will be removed and stored in a lens case, if required. | |
| 1.11. | Subjective sphero-<br>cylindrical refraction | Conduct a full spherocylindrical bare eye subjective refraction with binocular balance and record the resultant monocular visual acuity for each eye to the nearest letter. Note: The duo-chrome test should be used for refining the monocular and binocular spherical endpoints. This test will be considered to have reached the endpoint when the targets on red and green backgrounds appear to be equally sharp. However, if the subject's response changes immediately from "red" to "green" | |
| | | with a 0.25DS change in power, the endpoint will be<br>the most plus power (with "red" target clearer) before<br>this reversal. | |
| 1.12. | Slit lamp biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the visit will be discontinued; however, the subject may repeat the baseline evaluation (one time) at a later date once the condition lessens. Should the clearance of the fluorescein need to be expedited, preservative-free rewetting drops or artificial tears may be instilled. | |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.13. | Eligibility at baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. | _ |
| | | If subject is deemed to be ineligible after baseline, proceed to Final Evaluation. | |

| | | Visit 1: Lens Fitting # | 1 |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.14. | Lens selection | Assign the study lens based scheme. Select the fitting le corrected subjective refracts consideration of the following. 1. Label cylinder axis is rounding the refraction of degrees. Axis ending it rounded towards 180 frounded towards 180 frounded towards 180 frounded stigmatism, or towards frule astigmatism (e.g., 17 105 should be rounded to Cylinder power should be following table: | |
| | | Vertex corrected cylinder power (X) within the range: (DC) | |
| | | $-0.625 \le X < -1.125$ | $-0.625 \le X < -1.125$ $-0.75$ |
| | | $-1.125 \le X \le -1.625$ | -1.25 |
| | | 3. The fitting lens spherical (label sphere power + 1/2 power) should be as clos the vertex-corrected refravertex-corrected refraction between two label SE popower should be fit first. | |
| 1.15. | Right eye lens insertion | Instruct the subject to insert random orientation. | |
| | | If lens is uncomfortable, ins | |
| 1.16. | Timed rotation<br>assessments during<br>settling period | remove, reinsert, or replace as necessary. Start a stopwatch (or suitable smartphone or tablet timing app) as soon as the right lens is inserted. Record lens rotation (direction and magnitude) to the nearest degree at one (1) and three (3) minutes following insertion. | |
| | | Note: All lenses in this study have scribe marks at the 6 o'clock position and rotation measurements are made relative to a vertical reference line. | |

| | Visit 1: Lens Fitting #1 | |
|---|---|---|
| Step | Procedure | Details |
| 2000 - 1000 - 10 | | |
| 1.17. | Left eye lens insertion | Instruct the subject to insert the left-eye lens with random orientation. |
| | | If lens is uncomfortable, inspect for damage and |
| | | remove, reinsert, or replace as necessary. |
| 1.18. | Timed rotation | Start a stopwatch (or suitable smartphone or tablet |
| | assessments during | timing app) as soon as the left lens is inserted. Record |
| | settling period | lens rotation (direction and magnitude) to the nearest<br>degree at one (1) and three (3) minutes following |
| | | insertion. |
| | | Note: All lenses in this study have scribe marks at the |
| | | 6 o'clock position and rotation measurements are |
| 1.10 | T1" | made relative to a vertical reference line. |
| 1.19. | Lens settling | Allow lenses to settle until, in both eyes: Reflex tearing has subsided |
| | | The lens fit (centration and movement on blink) |
| | | has stabilized |
| | | The lens orientation has stabilized (orientation |
| | | scribe mark has reached it's settled position) |
| 1.20. | Toric fit assessment | Record for each eye: |
| | | The rotational position to the nearest degree |
| | | 2. Lens stability with blinks |
| | | Toric fit acceptability. The toric lens fit will be designated as 'unacceptable' if either: |
| | | a. The lens ABSOLUTE ROTATION is |
| | | greater than 20 degrees |
| | | b. The LENS STABILITY WITH BLINK is greater than 5 degrees |
| | | If one or both lenses demonstrate an unacceptable toric |
| | | fit, the subject will be discontinued (proceed to final |
| | | evaluation). |
| 1.21. | General lens fit | The fitting characteristics of the lens in both eyes will |
| | assessment | be assessed using a slit lamp. Lens position (centration, |
| | | limbal exposure, edge lift) and movement (primary and<br>up gaze as well as push-up) will be assessed. Fit |
| | | acceptability is defined as any lens that does <b>not</b> |
| | | display the following general fit characteristics: |
| | | Limbal exposure (presence of clear cornea) in |
| | | any direction of gaze. |
| | | Edge lift. |
| | | Insufficient movement in all three movement |
| | | assessments (primary gaze, up-gaze and push-up test). |
| | | Excessive movement in primary gaze. |
| | | If the general fit is unacceptable for either eye, the |
| | | subject will be discontinued (proceed to exit |
| | | evaluation). |

| | | Visit 1: Lens Fitting #1 | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | | <u> </u> |
| 1.22. | Spherical over-refraction | Perform monocular spherical over-refraction using duo-chrome to refine the endpoint as described in step 1.11 (the final spherical endpoint may be determined binocularly). | |
| | | The spherical over-refraction must be plano in both eyes to continue. | |
| | | If a non-plano over-refraction is found in either eye, the lens(es) must be refit with the indicated change in sphere power. If the indicated lens power is not available for either eye (e.g., outside the available SKU range), the subject will be discontinued (proceed | |
| 1.23. | Lens modification (if | to final evaluation). If modification is necessary in one or both eyes, select | g r |
| 1.23. | necessary) | the reason for refitting lenses: | |
| | | The settled lens rotation is such that a different cylinder axis would be more appropriate (use the LARS rule to determine the replacement lens cylinder axis) The spherical over-refraction is not plano Other (specify reason) Repeat steps 1.15 through 1.22 for one or both eyes, as appropriate. | |
| | | A maximum of 2 lens modifications are allowed per eye. If, for either eye, the fit is not successful after 2 modifications, the subject will be discontinued (proceed to final evaluation). | |
| 1.24. | Post-fit PRO questionnaire | Subjects will complete a PRO questionnaire regarding<br>the initial comfort, vision and handling of the study<br>lenses. | |
| 1.25. | Additional sample of<br>toric lens orientation (1) | Instruct the subject to leave the consulting room and walk around for at least 2 minutes. Upon their return, measure and record the toric lens orientation for each eye to the nearest degree. | |
| 1.26. | Additional sample of toric lens orientation (2) | Repeat the previous step once again. | |
| 1.27. | Exit visual acuity | Record the exit monocular distance Snellen visual acuity for each eye with the subject wearing the study lenses. | |
| 1.28. | Dispensing criteria | Lenses may be dispensed if both following conditions are met: 1. The monocular distance visual acuity with the study lenses is equal to or better than 20/25 in each eye. 2. The subject indicates that the comfort and vision with the study lenses is acceptable. If either of these conditions is not met, the subject will be discontinued (proceed to exit evaluation). | |
| 1.29. | Dispensing instructions | If the study lenses are suitable for dispensing: Minimum wear requirement: Instruct the subject to wear the study lenses for at least 8 hours per | |

| | Visit 1: Lens Fitting #1 | |
|---|---|---|
| Step | Procedure | Details |
| | | day (in a daily wear / daily disposable modality) on at least 5 days between the end of this visit and the start of the next visit. The day of the dispensing visit and/or the day of follow-up visit may be counted toward the 5 day requirement, but only if the study lenses are worn for at least 8 hours on those days. Note that, regardless of whether those days are counted toward meeting the minimum wear requirement, the return window requirement still holds (i.e., counting the day of this visit as day 0, the subject must still return for their next visit on day 5 through 9). |
| | | Subjects must not wear their habitual lenses at any time during study lens wear periods (spectacle wear is acceptable on non-wearing days). Provide the subject with a copy of the Patient Instruction Guide. |
| | | Preservative-free rewetting drops are permitted, if needed. |
| | | • Dispense enough lenses for the subject to complete the 14(±4) day wear period (i.e., up to and including the 2-week follow-up visit). At the investigator's discretion, in instances where there is a high likelihood of the subject needing replacement lenses (e.g., due to subject activities, unavailability of subject or site during the wear period, high likelihood of lens tears, etc.), additional pairs may be dispensed. |
| | | Note: In the event that a subject requires additional lenses due to loss or damage, they may return to the clinical site for lens replacement. As much as reasonably possible, damaged lenses and packaging should be returned to the clinical site (in solution, if possible) for shipping to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form, store the lens in a labeled vial with saline and return it to the Sponsor. |
| | | Ensure the subject is aware of the correct lens<br>power for each eye (label the lenses with R and L<br>as appropriate). |
| 1.30. | Schedule next visit | Schedule the next visit to occur in 7(±2) days (counting the day of this visit as day 0, the subject may return on day 5 through 9). Ensure the subject is instructed to wear the study lenses for at least 1 hour immediately prior to attending the next visit. |

#### VISIT 2

Visit 2 will occur 5 to 9 days following Visit 1. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

| | | Visit 2: Follow-Up # | 1 | | |
|---|---|---|---|---|---|
| Step | Procedure | Details | | | |
| 2.1. | Wear time and compliance | Record the subjects wearing time and comfortable wearing time. Subjects must have worn lenses for at least 8 hours on at least 5 days between the dispensing visit and this visit, and for at least 1 hour prior to attending this visit. | | | |
| 2.2. | Review medical history<br>and concomitant<br>medications | Record any changes to the<br>(including adverse events<br>medications. | | | |
| 2.3. | Subject reported ocular symptoms | Record any subject repor<br>response to a verbal oper<br>questionnaire. | | | |
| 2.4. | Follow-up PRO questionnaire | Subjects will complete a PRO questionnaire to assess their experience with the study lenses. The glare PRO questionnaire will be completed first, followed by the CLUE questionnaire, followed by the other PRO items. | | | |
| 2.5. | Entrance visual acuity | Record the entrance Snel wearing the study lenses. | | ch eye while | |
| 2.6. | Distance ETDRS visual acuity | Measure monocular discontrast (HLHC) visual 4 meters. Measure each eye using below: | acuity using E | TDRS charts | at |
| | | Condition | HI | HC | |
| | | Room illumination | > 40 | 0 lux | |
| | | Chart luminance | 120 - 20 | 00 cd/m <sup>2</sup> | |
| | | Eye | OD | os | |
| | | Charts | HC-1 | HC-2 | |
| 2.7. | Toric lens orientation | Recorded letter-by-letter results into EDC. Record the toric lens orientation for each eye to the nearest degree. | | | |
| 2.8. | Lens removal | Remove and place both lenses into a lens case with saline solution. Do not discard the lenses. | | | |

| Visit 2: Follow-Up #1 | | | |
|---|---|---|---|
| Step | Procedure | Details | <u></u> |
| 2.9. | Biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the subject must be discontinued, an adverse event will be recorded, and the subject will be monitored as per the guidelines given in section Error! Reference source not found Should the clearance of the fluorescein need to be expedited, preservative-free rewetting drops or artificial tears may be instilled. | |
| 2.10. | Reinsert study lenses | The subject will reinsert the study lenses they removed prior to biomicroscopy. | |
| 2.11. | Lens settling period | Following lens reinsertion, allow lenses to settle until, in both eyes: Reflex tearing has subsided The lens fit (centration and movement on blink) has stabilized The lens orientation has stabilized (orientation scribe mark has reached it's settled position) | |
| 2.12. | Exit visual acuity | Record the exit monocular distance Snellen visual acuity for each eye with the subject wearing the study lenses. | |
| 2.13. | Dispensing instructions | Provide the subject with additional study lenses (with the same lens code and power as dispensed earlier). • Minimum wear requirement: Instruct the subject to wear the study lenses for at least 8 hours per day (in a daily wear / daily disposable modality) on at least 5 days between the end of this visit and the start of the next visit. The day of the dispensing visit and/or the day of follow-up visit may be counted toward the 5 day requirement, but only if the study lenses are worn for at least 8 hours on those days. Note that, regardless of whether those days are counted toward meeting the minimum wear requirement, the return window requirement still holds (i.e., counting the day of this visit as day 0, the subject must still return for their next visit on day 5 through 9). | |
| | | <ul> <li>Subjects must not wear their habitual lenses at any time during study lens wear periods (spectacle wear is acceptable on non-wearing days).</li> <li>Preservative-free rewetting drops are permitted, if needed.</li> <li>Ensure the subject has enough remaining study lenses to complete the wear period through to the next follow-up visit (if additional lenses are needed, complete an unscheduled visit for lens resupply).</li> </ul> | |

| | Visit 2: Follow-Up #1 | |
|---|---|---|
| Step | Procedure | Details |
| | | Instruct the subject to bring their habitual spectacles or contact lenses to the next visit (to wear following removal of the study lenses). |
| | | Note: In the event that a subject requires additional lenses due to loss or damage, they may return to the clinical site for lens replacement. As much as reasonably possible, damaged lenses and packaging should be returned to the clinical site (in solution, if possible) for shipping to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form, store the lens in a labeled vial with saline and return it to the Sponsor. |
| | | <ul> <li>Ensure the subject is aware of the correct lens<br/>power for each eye (label the lenses with R and L<br/>as appropriate).</li> </ul> |
| 2.14. | Schedule next visit | Schedule the next visit (Visit 3) to occur in 7(±2) days (counting the day of this visit as day 0, the subject may return on day 5 through 9). Ensure the subject is instructed to wear the study lenses for at least 1 hour immediately prior to attending the next visit. |

#### VISIT 3

Visit 3 will occur 5 to 9 days following Visit 2. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

Subjects should bring their own habitual spectacles or contact lenses to this visit to wear following study lens removal.

| | Visit 3: Follow-Up #2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1. | Wear time and compliance | Record the subjects wearing time and comfortable wearing time. Subjects must have worn lenses for at least 8 hours on at least 5 days during the dispensing period, and for at least 1 hour prior to attending this visit. |
| 3.2. | Collect unworn lenses | Collect any unworn study lenses that were dispensed at the previous visit. |
| 3.3. | Review medical history<br>and concomitant<br>medications | Record any changes to the subject's medical history (including adverse events) or concomitant medications. |
| 3.4. | Subject reported ocular symptoms | Record any subject reported ocular symptoms in response to a verbal open-ended symptoms questionnaire. |

| Sirst, by the cts are |
|---|
| First,<br>y the |
| First,<br>y the |
| y the |
| y the |
| y the |
| rts are |
| ets are |
| in all |
| hile |
| they |
| e that |
| he<br>earing |
| euring |
| ile |
| he |
| and |
| turn,<br>he |
| ith |
| 1296 |
| py has |
| used to |
| as 3 or |
| adverse |
| nitored |
| erence |
| s 2 |
| to be |
| rtificial |
| on to |
| al |
| r |
| ng a |
| of this<br>rough |
| g the |
| <i>S</i> |
| reconstitution of the constitution of the cons |

#### VISIT 4

Visit 4 will occur 5 to 9 days following Visit 3. Subjects may wear their habitual contact lenses to this visit.

| | Visit 4: Continuance | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.1. | Review medical history<br>and concomitant<br>medications | Record any changes to the subject's medical history or concomitant medications. | |
| 4.2. | Subject reported ocular symptoms | Record any subject reported ocular symptoms in response to a verbal open-ended symptoms questionnaire. | |
| 4.3. | Entrance visual acuity | Record the entrance distance Snellen visual acuity for OD and OS with the subject wearing their habitual correction. | |
| 4.4. | Remove habitual lenses (if worn) | If worn, the subject's habitual contact lenses will be<br>removed. Lenses may be stored in a lens case, if<br>required. | |
| 4.5. | Biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the subject must be discontinued, an adverse event will be recorded and the subject will be monitored as per the guidelines given in section Error! Reference source not found. | |
| | | Should the clearance of the fluorescein need to be expedited, preservative free rewetting drops or artificial tears may be instilled. | |
| 4.6. | Continuance | Verify that the subject is eligible to continue in the study. | V<br>S |

#### Visit 4: Lens Fitting #2

The steps followed will be the same as those listed under Visit 1: Lens Fitting #1.

#### VISIT 5

Visit 5 will occur 5 to 9 days following Visit 4. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

#### Visit 5: Follow-Up #3

The steps followed will be the same as those listed under Visit 2: Follow-Up #1.

#### VISIT 6

Visit 6 will occur 5 to 9 days following Visit 5. Subjects must present to this visit wearing the study lenses in both eyes, and lenses must have been worn for at least 1 hour prior to the visit.

Subjects should bring their own habitual spectacles or contact lenses to this visit to wear following study lens removal.

| Visit 6: Follow-Up #4 | | |
|---|---|---|
| Step | Procedure | Details |
| 6.1. | Wear time and compliance | Record the subjects wearing time and comfortable wearing time. Subjects must have worn lenses for at least 8 hours on at least 5 days during the dispensing period, and for at least 1 hour prior to attending this visit. |
| 6.2. | Collect unworn lenses | Collect any unworn study lenses that were dispensed at the previous visit. |
| 6.3. | Review medical history<br>and concomitant<br>medications | Record any changes to the subject's medical history (including adverse events) or concomitant medications. |
| 6.4. | Subject reported ocular symptoms | Record any subject reported ocular symptoms in response to a verbal open-ended symptoms questionnaire. |
| 6.5. | Follow-up PRO<br>questionnaire | Subjects will complete a PRO questionnaire to assess their experience with the study lenses. |
| | | The glare PRO questionnaire will be completed first, followed by the CLUE questionnaire, then the other PRO items, then the preference questionnaire. |
| | | Note: within the glare PRO questionnaire, subjects are asked to compare their experiences with glare while using the study contact lenses against the lenses they wore just before starting the study. Please ensure that subjects understand that the comparator lens is the habitual brand of the contact lenses they were wearing prior to the study. |
| 6.6. | Entrance visual acuity | Record the entrance Snellen VA for each eye while wearing the study lenses. |
| 6.7. | Toric lens orientation | Record the toric lens orientation for each eye to the nearest degree. |
| 6.8. | Additional sample of toric lens orientation (1) | Instruct the subject to leave the consulting room and walk around for at least 2 minutes. Upon their return, measure and record the toric lens orientation to the nearest degree in each eye. |
| 6.9. | Additional sample of<br>toric lens orientation<br>(2) | Repeat the previous step once again. |
| 6.10. | Lens removal | Remove and place both lenses into a lens case with saline solution. Do not discard the lenses until after biomicroscopy has been completed. |
| Visit 6: Follow-Up #4 | | |
|---|---|---|
| Step | Procedure | Details |
| 6.11. | Biomicroscopy | The FDA Slit Lamp Classification Scale will be used to grade findings. If any slit lamp finding is graded as 3 or worse, the subject must be discontinued, an adverse event will be recorded, and the subject will be monitored as per the guidelines given in section Should the clearance of the fluorescein need to be expedited, preservative-free rewetting drops or artificial tears may be instilled. Study lenses may be discarded if there is no reason to store them following biomicroscopy. |

## FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Subject Disposition | Indicate if the subject completed the study successfully. If the subject is discontinued from the study, indicate the reason. |
| F.2 | Exit Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best-corrected distance visual acuity (OD and OS) to the nearest letter. Note: This step is not necessary if the subject was |
| | 7 | exited due to screen failure. |
| F.3 | Exit Slit Lamp<br>Biomicroscopy (for<br>subjects that are<br>discontinued early) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessary if the subject was exited due to screen failure. |
| | | Note: This step is not necessary if the subject was exited due to screen failure, or if biomicroscopy was performed as part of the final follow-up visit procedures (i.e., immediately prior to the final evaluation). |

# 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the
  adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.

- · Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pre-treatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | tep Procedure Details | |
| U.1 | Reason for unscheduled visit | Indicate if the <u>only</u> reason for the visit is that the subject requires additional test articles. If the reason is other than resupply of previously dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if applicable) | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.3 | Adverse Events and<br>Concomitant<br>Medications Review (if<br>applicable) | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.4 | Entrance VA (if applicable) | Record the entrance distance visual acuity (OD, OS) to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical Refraction (if<br>applicable) | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS). |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. |
| U.8 | Exit Visual Acuity (if applicable) | Record the subject's exit distance visual acuity (OD, OS) to the nearest letter. |

**NOTE**: If the only reason for the unscheduled visit is that the subject requires additional test articles, only the dispensing information needs to be recorded.

#### 7.4. Laboratory Procedures

Not applicable.

## 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- have not withdrawn/discontinued from the study for any reason described in section 8.2.
- completed all visits through the final visit (visit 6).
- If all visits were completed but an additional visit is considered necessary for subject care, follow the requirements for unscheduled visits in section 7.3.

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol.
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear.
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject misses any study visits.
- Subject not compliant with study lens wear schedule.
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation.

Additional subjects may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

## 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed concomitant interventions for this study include ocular medications of any kind, or any systemic medications that would normally contraindicate contact lens wear or may otherwise compromise study endpoints.

#### 9.1. Systemic Medications

Certain systemic medications are known to have a higher likelihood to interfere with contact lens wear, chiefly by disrupting the tear film.

A summary of disallowed systemic medications is shown in Table 4. Subjects with a history of taking these medications will be allowed to enroll only if:

- The medications have been taken on a continual, routine basis for at least 6 months, and
- The subject has demonstrated successful contact lens wear during this time.

Or:

The subject was taking the medication on a temporary basis and ceased taking that medication at least 2
weeks prior to signing the informed consent (this is considered sufficient time for the medication to have
left the body prior to enrollment).

Subjects with a history of taking medications listed in Table 4 on a long-term, routine basis for less than 6 months will not be allowed to participate in the study.

Table 4: Disallowed systemic medications

| Class of Drug Common Indication(s) | | Common Examples |
|---|---|---|
| Estrogens (not including contraceptive medication) | Menopause, osteoporosis, vaginitis | Vagifem, Estrace, Climara, Vivelle-Dot, Premarin, Minivelle, etc. |
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent, Hyosyne,<br>Levsin, Symax Fastab, Symax SL,<br>Homax SL, Cogentin, Transderm Scop,<br>etc. |
| Beta-blockers | Hypertension, angina, heart attack, migraine, artrial fibrillation, andrenal cancer, essential tumor, glaucoma | Toprol XL, Lopressor, Tenormin,<br>Propranolol, Timoptic, Trandate, Inderal<br>LA, etc. |
| Psychotropics | Antipsychotic (schizophrenia, mania),<br>antidepression, antiobsessive, antianxiety,<br>mood stabilizer, stimulants (ADHD) | Zoloft, Celexa, Prozac, Lexapro,<br>Effexor, Cymbalta, Ativan, Xanax,<br>Desyrel, Wellbutrin, etc. |
| Vitamin A analogs | | Isotretinoin |

Examples of disallowed systemic antihistamines are given in Table 5. Subjects with a history of taking systemic antihistamines will be allowed to enroll only if:

- . They have taken antihistamines continuously for at least 2 weeks, and
- · They have demonstrated successful wear while taking the medication

Or:

• They stopped taking the medication for at least 2 weeks prior to enrollment.

Table 5: Disallowed systemic antihistamines

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Antihistamines | Allergic rhinitis, sedation, hives, allergic conjunctivitis, skin allergy, itching, motion sickness | |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report

deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation." Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 6 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 6: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended > 3 days out of visit<br>window defined in study<br>procedures | Visit attended ≤ 3 days out of visit window defined in study procedures |
| Unanswered PRO questions | If questionnaire is not completed (i.e., all questions are unanswered) for any visit. | Any individual PRO questions are unanswered (i.e., left blank). |
| Insufficient wear of study lenses | Subject does not wear study lenses for at least 8 hours on at least 5 days of a study lens dispensing period. | Subject does not wear study lenses<br>for at least 1 hour prior to attending<br>a follow-up visit. |
| | Subject wears their habitual lenses<br>during any of the study lens wear<br>periods. | |

In the case of a major protocol deviation, the decision of whether or not the subject will be excluded from the Per-Protocol analysis population will be made at the time of cohort review.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.

• Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB." Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

**Serious Adverse Event (SAE)** – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect

• Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

**NOTE** 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device. **NOTE** 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

## 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e., the relationship between the test article, study treatment or study procedures, and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).

- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

#### 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g., concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g., concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g., concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g., it is confirmed by de-challenge and re-challenge.

## 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment, or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study, it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1. Reporting Adverse Events to Sponsor

Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

## **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None.

# 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

## 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

Descriptive statistics will be reported for all key variables as appropriate. Continuous data will be summarized descriptively by sample size (n), mean, standard deviation (SD), median, minimum (Min) and maximum (Max). Categorical data will be summarized descriptively by frequency count (n) and percentage (%) of subjects or eyes within each category level. Summary tables will be presented by event (Baseline, Fitting, 1-week follow-up, 2-week follow-up, Unscheduled and Final Evaluations) and study lens type (Test and Control) as applicable, for the analysis set of interest. The denominator for all percentages will be the number of subjects (or eyes as applicable) with available data in the lens group under consideration. Unscheduled visits and tele-visits will be summarized separately and will be excluded from the primary and secondary analysis.

All available data collected at scheduled visits will be used in the statistical summaries and analyses, with no imputation of missing data. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis. All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC).

# 14.2. Sample Size Justification

This study was not designed or powered to test any statistical hypotheses with respect to incidence (percentage) of study lens-related grade 3 or higher SLFs after approximately 2-weeks of lens wear. Instead, the sample size and study design were based on clinical considerations and operational feasibility. A sample size of 60 subjects (120 eyes) to complete (through Visit 6), will provide adequate precision around the estimate of the percentage of eyes with study lens related grade 3 or higher SLFs as measured by the half-width of a 95% CI. Percision estimates were provided using difference scenarios for the percentage of events and are displayed in Table 7 below.

Table 7: Half-Width of the 95% Confidence Intervals for Proportion of Eyes with Grade 3+ SLFs

| Sample Size (number of subject to complete) | Proportion of Grade 3 +<br>SLFs | Confidence Interval<br>Half-Width | Estimated Upper Limit |
|---|---|---|---|
| 60 (120 eyes) | 0 (no events) | 0.02466 | 0.02466 |
| | 0.0083 (1 event) | 0.03057 | 0.03887 |
| | 0.0167 (2 events) | 0.03488 | 0.05158 |

A total of 60 subjects are targeted to complete the study. To account for subject drop-out approximately 66 (based on a drop-out rate of 10%) subjects will be enrolled in this study to ensure that at least 60 subject complete the study.

# 14.3. Analysis Populations

## **Safety Population:**

All subjects who are administered at least one treatment (study lens). Subject will be analyzed per actual treatment received.

#### **Per-Protocol Population:**

All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification for the exclusion of subjects with protocol deviations from the per-protocol population set will be documented in a memo to file.

## **Intention-to-Treat (ITT) Population:**

All randomized subjects. Subject will be analyzed per planned randomized treatment.

#### 14.4. Level of Statistical Significance

Not applicable, there is no planned hypothesis testing for any endpoints in this study.

#### 14.5. Primary Analysis

The summary of the primary endpoint will be conducted on the safety population.

The distribution of eyes (n, %) with SLF grade level will be summarized by study lens type. The grading SLFs scale is from 0 to 4, where Grade 0 represents the absence of findings and 1 to 4 representing successively worse findings (i.e., Grade 1 = trace, Grade 2 = Mild, Grade 3 = moderate and Grade 4 = severe).

# 14.6. Secondary Analysis

Not applicable.

# 14.7. Exploratory Analyses

Summary for exploratory endpoints will be provided for both the ITT and the Per-Protocol populations. However, all analyses for exploratory endpoints will be conducted on the ITT population.

# Distance Monocular HLHC logMAR visual acuity

Distance monocular HLHC logMAR visual acuity at the 1-week follow-up will be summaried and presented only descriptively by lens type accompanied with the 2-sided 95% CIs. Summary statistics are described in section 14.1.

# CLUE Comfort, Vision, and Handling Scores

The analysis of exploratory endpoints of CLUE comfort, vision and handling at the fitting, 1-, and 2-week follow-up visits will be conducted separately for each CLUE domain. The exploratory analysis of each CLUE score endpoints will include the estimation of mean CLUE scores and associated 95% CIs for each study lens (Test lens and Control lens). Additionally, the mean difference between the Test and Control lens paired with the 95% CI will be calculated.

CLUE scores will be analyzed using a linear mixed model, adjusting for baseline scores as a covariate. Sequence of lens wear, study period, lens type (Test and Control), timepoint (fitting, 1-week, and 2-week follow-up visit), and the ineraction lens type by timepoint will be included as fixed effects. Other baseline characteristics such age, gender, and/or race will be included as fixed covariates when appropriate. Site and subject nested within site will be included as random effects (G-side). Residual errors from measurements within the same subject and timepoint across study period will be modeled using an unstructured covariance structure (UN). If the model does not converge, other covariance structures will be considered. The Kenward and Roger method will be used for the denominator degree of freedom. Estimates for each study lens and between study lenses (Test lens and Control lens) will be carried out using two-sided 95% CIs for the least-square mean and/or mean difference.

## Toric Lens Orientation

The distribution (counts, percentages) of eyes for the toric Orientation (in degrees) at 1- and 3-minutes after lens insertion will be summarized by timepoint (fitting, 1-, and 2-week follow-up) and lens type.

# Mean Settled Lens Orientation

Mean settled lens orientation will be summarized separately for each timepoint (fitting, 1-, and 2-week follow-up visits) and lens type (Test and Control). Mean settled lens orientation is calculated by eye by averaging across all lens orientation measurements collected at least 15-minutes after lens insertion. The standard deviation of average settled lens orientation will also be calculated.

The exploratory analysis of this exploratory endpoint will include the estimation of the mean settled rotation by study lens paired with the corresponding two-sided 95% CIs for each lens, and the point estimate with the two-sided 95% CI for the mean difference.

Mean settled rotation will be analyzed using a linear mixed model. Sequence of lens wear, period, lens type, and first order carryover effect will be included in the model as fixed effects. Other baseline characteristics may be included, such as, race and age. Subject will be included as a random effect. Residual errors between measurements within a subject across periods will be modeled using an unstructured (UN) covariance structure. The Kenward and Roger Method will be used for the calculation of denominator degrees of freedom. Estimates will be calculated using two-sided 95% confidence intervals constructed for the least-square mean and/or least-square mean difference.

#### Adverse Events

All Adverse Events reported during this study will be provided in a listing. This listing will include subject demographic information, treatment information (associated with the time of the reported AE), AE type (ocular or non-ocular), seriousness / classification, causality or relatedness, adverse event severity, outcome, actions taken and the associated start and end date / time for each AE.

Additional exploratory analyses may be considered at the discretion of the study sponsor.

#### 14.8. Interim Analysis

Not applicable.

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the Sitero EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

No external data sources will be included in this study.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the

Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

# 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov by the Sponsor.

# 16. DATA MANAGEMENT

## 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, including the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal

Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

## 16.4. Data Monitoring Committee (DMC)

Not applicable.

## 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test articles and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

## 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study, and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the subject is fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily.

### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, according to ISO 14155:2020¹ and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64th WMA General Assembly 2013² and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with ISO 14155:2020¹ and applicable regulatory requirements.

## 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects).
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The

informed consent is in accordance with principles that originated in the Declaration of Helsinki<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA)<sup>8</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor

personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

## 19. STUDY RECORD RETENTION

In compliance with the ISO 14155:2020,¹ the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ISO 14155:2020¹ and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports.

If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

## 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

# 21. PUBLICATION

There is no plan to publish the outcome of this investigation.

#### 22. REFERENCES

1. ISO 14155:2020: Clinical investigation of medical devices for human subjects — Good clinical practice, Available at: https://www.iso.org/standard/71690 html.

- 2. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects, Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 3. United States (US) Code of Federal Regulations (CFR). Ophthalmic Drug Products for over-the-counter human use, Section 349.1. Available at: https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?fr=349.1.
- 4. Straker B. *Investigator's Brochure CR-6553. (VIS-CSIB-006511). Daily disposable toric contact lenses manufactured in senofilcon A with a blue light-filtering chromophore.* October, 2023.
- 5. RJ Wirth, MC Edwards, Henderson M, et a. Development of the contact lens user experience: CLUE scales. . *Optometry and Vision Science*. 2016;93(8):801. Available at: https://pubmed.ncbi.nlm.nih.gov/27383257/
- 6. SAS Institute Inc: SAS® 9.4 Statements: Reference, Third Edition. Cary, NC SAS Institute Inc; 2014.
- 7. MG Kenward, Roger J. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics.* 1997;53(3):983. Available at: http://dx.doi.org/10.2307/2533558
- 8. Health Information Portability and Accountability Act (HIPAA), Available at https://www.hhs.gov/hipaa/for-professionals/privacy/index.html

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)





CR-6553, v3.0

PRO SPECIFICATION Version 4 Final 2023-11-09
Page 61 of 132

JJVC CONFIDENTIAL



CR-6553, v3.0



CR-6553, v3.0








16









## APPENDIX B: PATIENT INSTRUCTION GUIDE

A Patient Instruction Guide (PIG) will be provided separately.

| APPENDIX | C: PACKAGE | INSERT | (APPROVED | PRODUCT) |
|----------|------------|--------|-----------|----------|
| | | | | INODUCI |

Alcon DAILIES TOTAL1® for Astigmatism (delefilcon A) soft contact lenses for Daily Disposable Wear.

## Alcon

## Package Insert for Alcon DAILIES TOTAL1™ for Astigmatism (delefilcon A) soft contact lenses for daily disposable wear

W900409251

INFORTANT: This package insert is effective as of May 2020 and applicable to the deleticon A contact lenses described below. Please read carefully and keep this information for future use.
This package insert is intended for the fay Care Principles of the package in a promptive insert that principles in the Pather Instruction Bendetia to make what who who that page for carefully carefully appreciate the package insert and the Pather Instruction Bendetia are available whoth charges from cycling Continuer Service at 1-800-241-3998 or do ns that pertain to the patient's prescribed lenses. Alcon also recor -800-241-5999 or download from our website at www.alcon.com



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed Eye Care Professional.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1™ for Astigmatism (delefilcon A) soft contact lenses are made of a DIALLES UPIAL "To Assignation (celention 4) soft contact tenses are made or the lens material that is approximately 35% water and 67% (deleftion 4) polymer, a silicone containing hydrogel with added phosphatidy/choline. The core lens material containing 35% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copyer phthatiogranine, and have a light blue-green into that makes them easier to see when handling. This package insert applies to DAILLES TOTAL "Me for astignation lenses with light absorbing chromophores iss identified in "Contents" statement on carbon handles. Reported to Marcel 16% the absorbine precisions are seen seen seen seen to be for the handles. Reported to Marcel 16% the absorbine precisions are seen seen seen seen to be for the handles. Reported to Marcel 16% the absorbine precisions are seen to be for the handles. Reported to Marcel 16% the absorbine precisions are seen to the body the handless the content of the seen the seen seen seen to be the first the material to the seen that the seen that the seen that the seen that the seen that the seen that the material than the seen that the seen that the seen that the seen that the seen that the material than the seen that the radiation and reduce transmittance of high energy visible light (HEVL) wavelengths in the range from 380 nm to 450 nm\*.

Lens Properties
• Refractive Index (hydrated): 1.42

Light Transmittance

90% ± 5% for average over 380 to 780 nm ≤ 80%T at 420 nm (refer to Figure 1 for

transmittance profile)\*  $\tau$ UVB < 1.0 % (average percent transmittance over 280 nm to 315 nm) IN Transmittance:

 $\tau UVA < 10.0$  % (average percent transmittance over 315 nm to 380 nm)

140 barrer units, measured at 35 °C (intrinsic Dk -Coulometric method) · Oxygen Permeability (Dk):

33% by weight in normal saline . Water Content:

#### **Lens Parameters**

Diameter Range: 13.0 to 15.0 mm Power Range: -20.00 to +20.00 D . Base Curve Range: 8.0 to 9.2 mm

## DAILIES TOTAL 17th for Astigmatism (delefilcon A)

Chord Diameter: 14.5 mm 0.11 mm @ -3.00 D (varies with power) Center Thickness

 Sohere Power: +4.00 to -6.00 D (0.25 D steps): -6.50 to -8.00 D

 Cylinder Power: -0.75 D, -1.25 D, -1.75 D, -2.25 D 10° to 180°, in 10° steps

When hydrated and placed on the comea, DALLES TOTAL1™ for Astigmatism (delefficon A) soft contact lenses act as a refracting medium to focus light rays on

The lenses contain a combination of UV and UV-Vis blocking monomers to help The lenses contain a combination of UV and UV-Vis blocking monomers to help protoct against transmission of narmful UV radiation to the cornea and into the eye. For example, a lens with 0.09 mm center thiskness (-3.00 D, thinnest projected parameter) blocks 97% of UVA radiation, and 99% UVB radiation average across the spectrum. The lenses reduce high energy visible light (HEVL) radiation reaching the back of the eye by about 33% in the range from 380 mm to 450 mm. See Figure 1 for the transmittance profile of deliction of kenses with light absorbing chromophores (-3.00 D, thinnest projected parameter). The radiation transmittance will be further context with increasion lens the firement. will be further reduced with increasing lens thickness

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV WARNINE UV absorbing contact lenses are NOT substitutes to protective UV absorbing eyewers, such as UV absorbing poggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewers as directed. NOTE: Long-term exposure to UV realistion is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental

cataracts. Exposure is based on a number of factors such as environmental conditions faithtie, exporagin, found oversi and personal factors (setter and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical states have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. High energy visible light filtering provided by detellicon A soft contact lenses with light absorbing chromophores is additive to the natural crystalline lens. There is no demonstrated clinical benefit to a 33% reduction in visible light at weavelengths below 450 nm. The Eye Care Professional should be consulted for more information.

Figure 1 illustrates the transmittance of a lens with 0.09 mm center thickness (-3.00 D, thinnest projected parameter), a human comea, a human lens, and the combined filtration effect of the contact lens and the human lens on retinal exposure. The shader regions of the graph represent the integrated attenuation transmittance percentages of the deletition A lenses with light absorbing chromophores (-3.00 D, thinnest projected parameter) in the high energy visible light region (300 mm to 450 mm). The overall light attenuation over this region is 33%\*, with 65% attenuation over the region from 400 mm to 450 mm. This represents the filtration of the contact lens through the central 6 mm portion for a lens with 0.09 mm center thickness

(-3.00 D, thinnest projected parameter). Filtration would increase for contact lens powers with higher center thickness.

| Wavelength | Percent integrated attenuation<br>transmittance of high energy<br>visible light* |
|---|---|
| 380 nm to 400 nm | 65% |
| 400 nm to 450 nm | 21% |
| 380 nm to 450 nm | 33% |



- Delefilcon A with light absorbing chromophores: Contact lens with 0.09 mm center thickness measured through central 6 mm portion for the
- thinnest marketed lens (-3.00 D, thinnest projected parameter). Human Cornea from a 24 year old person as described in Lerman S., Radiant Energy and the Eye, MacMillian, New York, 1980, p.58, Figure
- Human crystalline lens from a 25 year old person as described in Waxler M., Hitchins V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, Figure 5.
- Combined filtering effect of the contact lens and the natural crystalline lens

nure 1: Transmittance of a DAILIES TOTAL 1<sup>th</sup> for Astigmatism (delefik ntact Lens versus a Human Cornea and a Human Crystalline Lens

DAILIES TOTAL1™ for Astigmatism (deleflicon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to 6.00 diopters (D) of astigmatism.

The lenses are to be used for single use, daily disposable wear (less than 24 hours while awake) only. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

#### CONTRAINDICATIONS (Re

#### DO NOT use delefilcon A soft contact lenses when any of the following exists:

- Microbial infection of the eye Inflammation or infection of the anterior chamber of the eve
- Any active disease, injury, or abnormality affecting the comea, conjunctiva, or eyelids that may be exacerbated by contact lens wear
- Inadequate tear film (dry eye) that interferes with contact lens wear Reduced corneal sensitivity (corneal hypoesthesia)
- If eyes become red or irritated
- Use of any medication that is contraindicated or interferes with contact lens wear, including certain eye medications
- Any systemic disease which may be exacerbated by or interferes with safe contact lens wear, handling, or care
- Allergic reactions of the ocular surfaces or adnexa that may be caused by or exacerbated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance, or abnormal ocular response to contact lens

#### WARNINGS

#### Advise patients of the following warnings pertaining to contact lens wear:

- Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their Eye Care Professionals directions and all labelling instructions for proper use of lenses and lens care products. Eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.
- It a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her Eye Care Professional. It is recommended that contact lens wearers see their Eye Care Professional regularly as directed.
- Studies have shown that contact lens wearers who smoke have a great suffering ulcerative keratitis than among those who are nonsmokers.
- Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results' have shown that the risk of ulcerative keratitis is greater for daily wear users who wear their

- lenses overnight (outside the approved indication) compared to those who do not wear them overnight.

  Non-sterile liquids (i.e., tap water, distilled water, homemade saline solution, or
- saliva) should not be used as a substitute for any component in the lens care process. The use of tap and distilled water has been associated with Acanthamoeba keratitis, a comeal infection that is resistant to treatment and

#### PRECAUTIONS

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

#### Special Precautions for the Eve Care Professional

The following patients may not be suitable candidates and/or may experience a higher rate of adverse effects associated with contact lens wear:

- Patients with a history of non-compliance with contact lens care and disinfection regimen, wearing restrictions, wearing schedule or follow-up visit schedule.
- Patients who are unable or unwilling to understand or comply with any ravens who are unable or unwining to understand or comply with and directions, warnings, precations, or restrictions. Contributing stactors may include but are not limited to age, infirmity, other mental or physical conditions, and adverse working or living conditions.

  Patients with diabetes may have reduced corneal sensitivity. As a result, they are more prone to corneal injury and will not heal as quickly or completely as non-diabetics.

Note regarding lens designs and parameters:

Due to the small number of patients enrolled in the clinical investigation of Due to the smail number or patients erroried in the clinical investigation or lenses, all fractive powers, design configurations, and lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness, and optic zone diameter

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction. Therefore, the conflusing ocular health of the patient and less performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing Eve Care Professional.

Note the following precautions during initial dispensing and subsequent visits:

- ote the following precautions during initial dispensing and subsequent visits: Pluresceid, a yellow dys, should not be used while the lenses are not the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in-eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye.
- Instruct the patient to remove the lenses immediately if the eye becomes red or
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.
- Patients who wear contact lenses to correct prestypopia may not achieve the best corrected visual acuity for either far or near vision. Vision requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the Eye Care Professional's office, patients should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.

## Eye Care Professionals should carefully instruct the patient to take the following care regimen and safety precautions:

- Be sure that before leaving the Eye Care Professional's office, the patient is able to promptly remove lenses or have someone else available to remove them.
- Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse, and dry hands with a lint-free towel before handling lenses.
- Carefully follow the handling, insertion, removal, cleaning, dininfecting, storing, and wearing instructions in the Patient instruction Booklet for DAILIES TOTAL.17 for Astigmatism (delefilion A) Soft Contact Lenses and any additional instructions provided by the Eve Care Professional.
- Note the correct lens power for each eye to prevent getting them mixed up. Never use tweezers or other sharp objects such as fingernalls to remove lenses from the lens container.
- Always handle lenses carefully. If a lens is dropped, small particles or fibers may adhere to the lens surface, which can irritate the eye. Replace with a sterile new
- . Discard any lens that has become dehydrated or damaged. Replace with a sterile

#### Lens Wearing Precautions

- Remove the lenses before sleeping. Never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- Always keep a supply of replacement lenses on hand or have back-up spectacles available, as lenses should not be reused.
- Do not share lenses with anyone as this may spread microorganisms, which could result in serious eye health problems.
- Lenses should be disposed of each day upon removal from the eye. The lens should move freely on the eye at all times. If the lens sticks moving) on the eye, follow the recommended directions in the CARE FOR A STICKING, TORN, DRY, OR DECENTERED LENS section. If non-movement of the lens continues, consult your Eye Care Professional immediately.

<sup>\*</sup> See \*Note\*. There is no demonstrated clinical benefit to a 33% reduction in visible light at wavelengths below 450 nm.

- REMOVE THE LENS IMMEDIATELY if your eye becomes red or initiated.
- Promptly remove the lens to avoid serious injury in the event that dust, a foreign body, or other contaminant gets between the lens and the eye.
- Avoid all harmful or irritating vapors and furnes while wearing lenses to reduce the chance of lens contamination or physical trauma to the eye.
- Eye irritation, infection, or lens damage may result if cosmetics, lotion, soap, cream, hair spray, deodorant, aerosol products, or foreign particles come in contact with lenses. If sprays are used, eyes should be kept closed until the spray has settled.
- Consult an Eye Care Professional about wearing lenses during water sports and water related activities. Contact lens exposure to non-sterile water during activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection including, but not limited to, *Acanthamoeba* keratitis.
- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eve damage
- Do not use lenses beyond the expiration date.

#### Solution Precautions

Do not use saliva or any liquid other than the recommended solution for lubricating or rewetting drops with the lenses.

#### Other Topics to Discuss with Patients

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their Eye Care Professional at least once each year or as recommended by the Eye Care Professional.
- read titue each year to a recommend by the cyc during for tribescalar, Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, blurred vision, or visional changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquitizers, and those for motion sickness. Caution patients using these medications accordingly and prescribe proper remedial measures
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL1<sup>TM</sup> for Astigmatism (delefticon A) soft contact lens Patient instruction Booklet available from Alcon. It is important that patients understand its contents prior to

#### Who Should Know the Patient is Wearing Contact Lenses

- Instruct patients to inform their employers that they are wearing contact lenses Some jobs may require the use of eye protection equipment or may prohibit the wearing of contact lenses.
- Instruct the patients to inform their health care professionals that they are wearing contact lenses, as certain medications may interfere with contact

#### WATER ACTIVITIES

## Do not expose contact lenses to water while wearing them.

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when showering or swimming, discard them and replace with a new pair. Ask the Eye Care Professional for recommendations about wearing lenses during any activity involving water.

#### ADVERSE EFFECTS (Possible Problems)

Patients should be instructed to check their eyes regularly to make sure they look well, feel comfortable, and vision is clear.

Potentially serious complications are usually accompanied by one or more of the following signs and symptoms:

- Moderate to severe eye pain not relieved by removing the lens
- Feeling of something in the eye (foreign body sensation)
- Excessive watering or other eye secretions, including mucopurulent discharge
- Redness of the eyes
- Sensitivity to light (photophobia)
- · Burning, stinging, itching or other pain associated with the eyes
- t is less compared to when the lens was first placed on eye · Reduced sharpness of vision (poor visual acuity)
- · Blurred vision, rainbows, or halos around object
- · Feeling of dryness

mptoms, if ignored, may lead to more serious complications. These syr

#### WHAT TO DO IF A PROBLEM OCCURS

- If any of the above signs or symptoms occur:

  IMMEDIATELY REMOVE THE LENSES.
- . If the discomfort or problem stops, discard the lens and replace it with a new
- . If the discomfort or problem continues after removing the lens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) and contact an Eye Care Professional for Identification of the problem and prompt treatment to aw serious eye damage.
- Eve Care Professionals should inform the patient that a serious condition such as To call of trousous as anotous inform of peternic max a serious continuous con-comeal uicer, uicerative keratitis, infection, comeal vascualrazation, or insulti- as be present. These conditions may progress rapidly and may lead to permanent loss of vision. Less serious reactions such as a brasions, infiltrates, and bacterial conjunctivitis must be managed and treated properly to avoid more serious
- compications.

  Additionally, contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include, but are not limited to, local or generalized comeal edema, epithelial microcysts, epithelial straining, infiltrates, evoracusdirazion, endothelial polymegathism, tarsal papillary changes, conjunctival injection, or irtits.

## CARE FOR A STICKING, TORN, DECENTERED, OR DRY LENS

Patients should be informed that it may be possible to resolve less serious problems associated with contact tens wear by following the directions below. However, if following these directions does not resolve the problem, patients should consult their

towards unsecured and the control of

lens begins to move freely on the eye before attempting to remove it. It is important that you wash and dry your hands thoroughly before removing the lens. If the lens continues to stick, IMMEDIATELY consult your Eye Care

- It a lens tears in your eye, remove the pieces carefully by pinching them as you would for normal lens removal. If the lens pieces do not seem to remove easily, do not pinch the eye tissue. Rinse with sailer. If this does not help, contact the Eye Care Professional for assistance.
- If a lens decenters on the eye, it may be possible to re-center it by:
  - o Closing your eyelids and gently massaging the lens into place, or
  - o Looking in the direction of the lens and blinking gently, or
  - Gently pushing the off-centered lens onto the comea with light finger pressure on the edge of the upper or lower eyelid.
- Occasional dryness may be relieved by blinking fully several times or by the use of contact lens rewetting drops that are approved for use with soft contact lenses. If dryness persists, consult your Eye Care Professional.

#### **EMERGENCIES**

If chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes:

- · Flush eyes immediately with fresh saline solution or tap water
- Remove and discard lenses and immediately contact the Eye Care Professional or visit a hospital emergency room without delay.

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of delefficon A contact lenses, please notify: Alcon Medical Affairs in the USA at

#### FITTING GUIDE AND PATIENT ROOK! FT

Conventional methods of fitting contact lenses apply to DAILIES TOTAL1™ for Astigmatism (delefilicon A) contact lenses. For a detailed description of the fitting techniques, refer to the DAILIES TOTAL1™ for Astigmatism (delefilicon A) soft contact techniques, teler to the DALLES TOTAL "For Assignmation (periodical) soft the lens Professional Ritting and Information Guide or more information. Both the Professional Ritting and Information Guide and a Patient Instruction Booklet a available free of charge from:

Alcon Laboratories, Inc.

Fort Worth, TX 76134-2099, USA

or by calling Alcon Customer Service in the USA at:

## LENS WEAR AND REPLACEMENT SCHEDULE

- Daily Wear (less than 24 hours, while awake)

  Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24-hour period; however, optimum individual wearing schedules will vary.
- The maximum daily wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition because individual responses to contact lenses vary.
- Daily wear patients may initially over-wear the lenses. Avoid this tendency by carry was patients any initially over the little to a recommendative or stressing the importance of adhering to a proper initial wearing schedule. For patients who are new to daily wear, gradually increasing scheduled wearing time may allow ocular tissues to more easily adapt to contact lens wear.

#### Lens Replacement

Delefficon A contact lenses are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

#### LENS HANDLING INSTRUCTIONS

- Always wash and rinse hands thoroughly and dry completely with a clean, lint -free towel before handling contact lenses.
- Note the correct lens power for each eye to avoid getting them mixed up.
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination, which can lead to a serious eye infection.
- Shake the blister pack (containing a fresh new lens) gently prior to opening
- Remove the lens from the blister pack by carefully pouring it onto the palm of the
- Ensure that the lens is right side out.
- Inspect the lenses prior to insertion. Do not insert damaged or unclean lenses.
   Lens Insertion Instructions

- Wash and rinse hands thoroughly and dry completely with a clean lint-free
- Place a lens on the tip of your clean and dry right or left index finger. Place the middle finger of the same hand close to lower eyelashes and pull down the lower
- Use the fingers of the other hand to lift the upper eyelid.
- Place the lens directly on the eye (cornea) and gently roll finger away from the
- Look down and slowly release the lower lid.
- Look straight ahead and slowly release the upper lid.
- Blink gently.

## Lens Removal Instructions

- Wash and rinse hands thoroughly, and dry completely with a clean, lint-free
- Blink fully several times.
- While looking up, use the tip of the finger to slide the lens down onto the white part of the eye.
- Remove the lens by pinching gently between thumb and forefinger. Do not pinch the eve tissue
- If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance
- Never use tweezers or other sharp objects such as fingernals to remove lenses

## LENS CARE DIRECTIONS

- To help avoid serious eye injury from contamination, the Eye Care Professional should review the following instructions with the patient:
  Cleaning and disinfection of daily disposable lenses is not recommended. The

patient should be reminded to have replacement lenses or back-up spectacles available at all times.

Do not use saliva, tap water, homemade saline solution, distilled water, or ng other than the recommended rewetting drops or lubricants indicated for

#### DISPOSAL AND RECYCLING

Dispose of contact lenses and the blister pack lidding in the waste bin, not down the toilet or sink. The carton packaging and the polypropytene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste ment guidance

#### IN OFFICE USE OF TRIAL LENSES

The CHAIL USE OF THIS LEARNES EYE CAIP Professionals should educate contact lens technicians concerning proper use of trial lenses. Each contact lens is shipped sterile in a bifster pack containing phosphate bufferd saline southor. Hands should be thoroughly washer, inteed, and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the blister pack should not be opened until immediately prior to use. For fitting and diagnostic purposes, the lenses should be disposed of after a single use and not be re-used from patient to patient.

#### HOW SUPPLIED

Each lens is packaged in a foil-sealed plastic blister pack containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents outered sains solution with approximately 0.3% or polymenc wetting agents consisting of coopymers of polymenisomenie and polygracylamide-accylic) acid and is steam sterilized The package is marked with the base curve, diameter, dioptric power, oylhider axis and power (where applicable), ADD power (where applicable), manufacturing of number, date of manufacture, and appraish ordet. Lenses are supplied in cartons containing up to 90 individually sealed contact lenses.

#### The following may appear on labels or cartons:

| Symbol / Abbreviation | Description |
|---|---|
| BC | Base Curve |
| DIA | Diameter |
| PWR | Power |
| D | Diopter |
| L | Left |
| R | Right |
| CYL AXIS | Cylinder power and axis |
| UV | Ultra-violet |
| UVA | Ultra-violet A |
| UVB | Ultra-violet B |
| UV-Vis | Ultra-violet and Visible |
| HEVL | High Energy Visible Light (blue light) |
| 0 | Packaging waste license sign |
| 2 | Do not re-use |
| LOT | Batch code |
| ⊒ <sub>Exp</sub> | Use-by date<br>(Expiry date) |
| 0 | Single sterile barrier system |
| STERRED | Sterilized using steam |
| CE | European conformity mark |
| <b>en</b> | English (example of two letter code for the language) |
| Δ | Caution |
| | Consult instructions for use |
| <b>©</b> | Do not use if blister package is damaged |
| (8) | DO NOT DISPOSE LENSES IN TOILET OR SINK |
| _ | Manufacturer |
| ed . | Date of manufacture |
| MD | Medical device |
| | Authorized representative in the European Community |
| (B) ordy | CAUTION: Federal (United States) law restricts this devi-<br>to sale by or on the order of a licensed eye care profession |

#### Date: August 2021

Manufacturer: Alcon Laboratories, Inc. Fort Worth, TX 76134-2099, USA

 Check for actual product availability which may change over time.
 Cutter GR, Chalmers RL, Roseman M. The Clinical Presentation, Prevalence, and Risk Factors of Focal Corneal Infiltrates in Soft Contact Lens Wearers. The CLAO Journal Jan 1996: 22 (1): 30-37.

Schein OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Kenatitis Among Users of Daily-Wear and Extended-Wear Soft Contact Lenses The New England Journal of Medicine. 1989; 321(12):773-783.

## Alcon

© 2021 Alcon Inc.

W900409251-0821

# APPENDIX D: LENS FITTING CHARACTERISTICS SUBJECT REPORTED OCULAR SYMPTOMS DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS BIOMICROSCOPY SCALE DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION TORIC FIT EVALUATION DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE PATIENT REPORTED OUTCOMES LENS INSERTION AND REMOVAL VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING





| Title: | Lens Fitting Characteristics | |
|-----------------|------------------------------|--------------------|
| Document Type: | | |
| Document Number | . ' | Revision Number: 6 |





DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS










Title: **Biomicroscopy Scale Document Type: Document Number:** Revision Number: 10










**Document Type:** 

Document Number: Revision Number: 7



**Document Type:** 

Document Number: Revision Number: 7





| Title: | Toric Fit I | <b>Evaluation</b> | n |
|---|---|---|---|
| <b>Document Type:</b> | | | |
| <b>Document Number:</b> | | | Revision Number: 7 |



DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE







| Title:<br>Document Type: | Patient Reported Outcomes | | |
|--------------------------|---------------------------|------------------|----|
| <b>Document Number:</b> | | Revision Number: | 3 |
| | | 2 | |
| | | | a. |
| 0.00 | | | |



VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

| Title: | Visual Acuity Chart Luminance and Room Illumination Testing | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 4 |



#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6553 Evaluation of Delefilcon A and Senofilcon A Daily Disposable Toric Soft Contact Lenses Over Two Weeks of Wear

Version and Date: 3.0 27 November 2023

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020,¹ the Declaration of Helsinki,² United States (US) Code of Federal Regulations (CFR),³ and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |
